CLINICAL TRIAL: NCT07320690
Title: A Randomized Controlled Clinical Study of De-Escalation Surgery Following Immunotherapy for Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: De-Escalation Surgery After Immunotherapy in Locally Advanced Head and Neck Squamous Cell Carcinoma
Acronym: Neo-Margin
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Yue He, MD, Director of Oral and Maxillofacial & Head and Neck Oncology Department , Principal Investigator, Clinical Professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JYKQ-2025-057; NCRCO2025ZD-01 (Other Grant/Funding Number: Shanghai Ninth Peolple's Hospital)
Record Dates: First submitted 2025-11-29; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Head and Neck Squamous Cell Carcinoma; Locally advanced; De-escalation surgery; Standard surgery; Immunotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 to downgraded surgery (experimental) or standard surgery (control).
Masking Description: Open-label study; no parties are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- De-escalation surgery (Experimental): The surgical procedure should be designed and performed based on the tumor boundaries following neoadjuvant therapy.
  Interventions: Procedure: De-escalation surgery; Radiation: radiotherapy; Drug: adjuvant immunotherapy
- Standard Surgery (Active Comparator): The surgical procedure should be designed and performed based on the tumor boundaries prior to neoadjuvant therapy.
  Interventions: Procedure: Standard Surgery; Radiation: radiotherapy; Drug: adjuvant immunotherapy

INTERVENTIONS:
Procedure: De-escalation surgery — Surgical planning and resection will be conducted based on tumor boundaries assessed after neoadjuvant therapy.
  Arms: De-escalation surgery
Procedure: Standard Surgery — Surgical planning and resection will be conducted based on tumor boundaries assessed prior to neoadjuvant therapy.
  Arms: Standard Surgery
Radiation: radiotherapy — Radiotherapy is recommended within 6 weeks after surgery. Patients achieving a pathological complete response (pCR) may be exempted. For the primary tumor and involved nodes, 60-70 Gy in 30-35 fractions is delivered once daily, Monday to Friday (low risk: 60 Gy; high risk: 66 Gy; residual disease: 70 Gy). Suspected subclinical areas receive 45-50 Gy (2 Gy/f) or 54-63 Gy (1.6-1.8 Gy/f). Concurrent cisplatin is given when extracapsular nodal extension or positive/close margins (<1 mm) are present: 100 mg/m² every 3 weeks ×3, with renal function-based dose adjustment. For patients unsuitable for cisplatin, cetuximab is administered at 400 mg/m² in the first week, then 250 mg/m² weekly.
Drug: adjuvant immunotherapy — Postoperative adjuvant immunotherapy was administered in accordance with the initial treatment plan and clinical indications.
  Other Names: postoperative adjuvant immunotherapy

SUMMARY:
This is a multicenter, randomized, open-label, non-inferiority clinical trial designed to evaluate whether downgraded surgery-guided by post-immunotherapy tumor boundaries-can achieve comparable 3-year overall survival (OS) to standard surgery in patients with Stage III-IVa locally advanced head and neck squamous cell carcinoma (HNSCC) who have responded to neoadjuvant immunotherapy. A total of 356 patients will be randomized 1:1 to receive either downgraded or standard surgery, followed by risk-adapted adjuvant therapy. The primary endpoint is 3-year OS, with secondary endpoints including disease-free survival, quality of life, complication rates, and cost-effectiveness. The study hypothesizes that downgraded surgery will preserve organ function and quality of life without compromising survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years inclusive, with no restriction on gender.
2. Histologically confirmed primary squamous cell carcinoma of the head and neck (excluding nasopharyngeal carcinoma).
3. Clinical stage III-IVa according to the AJCC 8th edition TNM staging system prior to immunotherapy; specifically, stage III-IVa for oropharyngeal squamous cell carcinoma (p16-negative) or stage III for oropharyngeal squamous cell carcinoma (p16-positive).
4. ECOG performance status of 0 or 1.
5. Life expectancy of ≥6 months.
6. Received preoperative immune checkpoint inhibitor therapy, primarily with anti-PD-1 monoclonal antibodies or bispecific antibodies containing an anti-PD-1 arm, regardless of brand, with or without concurrent chemotherapy or targeted therapy, for no more than six cycles.
7. Achieved complete response (CR) or partial response (PR) on imaging assessment after preoperative therapy, according to RECIST 1.1 criteria.
8. Assessed as eligible for de-escalation surgery based on clinical evaluation by the surgeon. Examples include omission of surgery on the primary lesion; preservation of critical structures or functions, such as retaining the mandible initially planned for resection; avoidance of flap reconstruction; or limitation of tongue resection to less than half when hemi-glossectomy was initially indicated.
9. No prior curative surgery or radiotherapy for the current tumor.
10. Willing to undergo surgical treatment.
11. No significant contraindications to surgery.
12. Voluntary participation in the study, signed informed consent, good compliance, and willingness to cooperate with follow-up visits.

Exclusion Criteria:

1. Severe underlying diseases making the patient unable to tolerate surgery.
2. Current tumor is recurrent.
3. Myocardial infarction, severe/unstable angina, NYHA class II or higher heart failure, or symptomatic congestive heart failure within 6 months before randomization.
4. History of psychiatric drug abuse or drug addiction.
5. Pregnant or breastfeeding women.
6. Diagnosis of other malignancies within 5 years prior to study entry, except for locally treated and cured basal cell carcinoma or squamous cell carcinoma of the skin, superficial bladder carcinoma, carcinoma in situ of the cervix, ductal carcinoma in situ of the breast, and papillary thyroid carcinoma.
7. Any other severe physical or mental illness, or laboratory abnormalities that might increase the risk associated with participation or interfere with the study results, or any other conditions deemed unsuitable for participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2031-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival (OS) rate | 3 years
  The proportion of subjects in the intention-to-treat population who are alive at 3 years after randomization.

SECONDARY OUTCOMES:
5-year overall survival (OS) rate | 5 years
  The proportion of subjects in the intention-to-treat population who are alive at 5 years after randomization.
3-year and 5-year Event-free survival (EFS) rates | 5 years
  The proportion of subjects in the intention-to-treat population who have not experienced any EFS events at 3 and 5 years after randomization. EFS time is defined as the duration from randomization to the first occurrence of any of the following events: (1) disease recurrence or metastasis in patients who underwent surgery; (2) disease progression per RECIST 1.1, or recurrence/metastasis after non-surgical treatment (e.g., radiotherapy) following neoadjuvant therapy; (3) occurrence of a second primary tumor; or (4) death from any cause. Patients who did not undergo surgery due to clinical complete response (CR) or near CR, as well as those who declined surgery but received other antitumor therapies without experiencing progression, recurrence/metastasis, or death, or who had positive surgical margins without radiographic evidence of progression, are not considered to have reached an EFS event.
incidence of adverse events | Through study completion, an average of 5 years
  Adverse events observed will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Surgical complications | Perioperative
  Surgical complications in this study will be assessed according to the Clavien-Dindo classification system, and detailed information on all complications occurring during the perioperative period will be recorded in the eCRF.
Totally quality of life, QoL | Baseline, 1 months (±7d) after surgery and prior to radiotherapy, 2 months after radiotherapy, and 6 months (±14d) after randomization, 1year (±14d) after randomization
  Totally Health status and quality of life will be assessed using the European Organization for Research and Treatment of Cancer Quality of Lifer Questionnaire Core 30 (EORTC QLQ-C30) questionnaires.
Quality of life for HNSCC patients | Baseline, 1 months (±7d) after surgery and prior to radiotherapy, 2 months after radiotherapy, and 6 months (±14d) after randomization, 1year (±14d) after randomization
  Health status and quality of life will be assessed using the European Organization for Research and Treatment of Cancer Quality of Lifer Questionnaire Head and Neck 35 (EORTC QLQ-H&N35) questionnaires

OTHER OUTCOMES:
Pathologic complete response rate | Through study completion, an average of 5 years
  The proportion of patients who achieved pCR among the ITT population and the pathologically evaluable population in each group.
Major pathologic response rate | Through study completion, an average of 5 years
  The proportion of patients who achieved MPR among the ITT population and the pathologically evaluable population in each group.
Surgical resection rates stratified by anatomical subsite and extent of surgical downgrading | Through study completion, an average of 5 years
  The proportion of patients who received that level of surgery among those initially planned for surgical intervention at the corresponding subsite.
Primary tumor surgery exemption rate | Through study completion, an average of 5 years
  The proportion of patients who were exempted from primary tumor surgery among the ITT population in that group.
Lymph node dissection exemption rate | Through study completion, an average of 5 years
  The proportion of participants spared lymph node dissection among those originally planned for the procedure.
Blood loss volume | Intraoperative
  Intraoperative blood loss volume
Blood transfusion volume | Intraoperative
  Intraoperative blood transfusion volume
Tracheostomy rate | Through study completion, an average of 5 years
  The proportion of patients who underwent tracheostomy among the ITT population in that group.
Surgical mortality rate | Through study completion, an average of 5 years
  The proportion of patients who died from any cause within 28 days after surgery among the ITT population in that group.
Flap reconstruction exemption rate | Through study completion, an average of 5 years
  The proportion of patients exempted from free flap reconstruction among those who were initially planned to undergo the procedure within the group.
Length of hospital stay | Through study completion, an average of 5 years
  Total length of hospital stay was calculated from the day of surgery to the day of discharge (a stay of less than 24 hours was counted as 0.5 day). For patients who did not undergo surgery, the hospital stay was recorded as 0 days.
Inpatient surgical costs and radiotherapy/chemotherapy costs | Through study completion, an average of 5 years
  Medical costs incurred during the hospitalization for surgery and during postoperative radiotherapy and chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth Peolple's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No